CLINICAL TRIAL: NCT01335971
Title: Enhancing Nrf2 by Sulforaphane Treatment in COPD
Brief Title: Broccoli Sprout Extracts Trial to See if NRF2 is Enhanced by Sulforaphane Treatment in Patients With COPD
Acronym: BEST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Temple University (Other); State University of New York at Buffalo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1U01HL105569 (NIH); RFA-HL-10-003 (Other: NHLBI); NCT01318603 (obsolete NCT alias)
Record Dates: First submitted 2011-04-08; First posted 2011-04-15 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: COPD
Keywords: COPD; Nrf2; Sulforaphane
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sulforaphane 25 (Active Comparator): 25 micromoles (4.4 mg) sulforaphane daily by mouth
  Interventions: Drug: Sulforaphane 25
- Sulforaphane 150 (Active Comparator): 150 micromoles (26.6 mg) sulforaphane daily by mouth
  Interventions: Dietary Supplement: Sulforaphane 150
- Placebo (Placebo Comparator): Microcrystalline cellulose
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sulforaphane 25 — 25 micromoles (4.4 mg) sulforaphane daily by mouth
  Other Names: This is derived from broccoli sprouts.
  Arms: Sulforaphane 25
Dietary Supplement: Sulforaphane 150 — 150 micromoles (26.6 mg) sulforaphane daily by mouth
  Arms: Sulforaphane 150
Other: Placebo — Microcrystalline cellulose once daily by mouth
  Arms: Placebo

SUMMARY:
Evidence from investigators' group has shown that chronic obstructive pulmonary disease (COPD) patients have impairment of antioxidant defenses which are caused by a defect in activity of Nrf2. This trial focuses on sulforaphane, a derivative of cruciferous vegetables, which is a potent stimulator of Nrf2 activity. The investigators want to investigate whether ingestion of sulforaphane by COPD patients will increase Nrf2 activity and expression of downstream antioxidants. Accordingly, the investigators are conducting a placebo-controlled randomized proof of principle trial of two oral doses of sulforaphane, 25 and 150 micromoles, for 4 weeks in 90 COPD patients. The investigators' goal is to establish a safe and tolerable dose of sulforaphane that effects in vivo antioxidants via Nrf2, then the investigators will have a novel candidate treatment for longer-term efficacy trials.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a major cause of morbidity and mortality in the United States and is a growing cause of chronic disease internationally. Presently, there are limited treatment options for this disease to modify the progression of airflow obstruction and decrease periodic exacerbations. Recent evidence has emphasized the central role of oxidative stress as a mechanism of COPD pathobiology. Evidence from investigators' group has shown that COPD patients and animals exposed to cigarette smoke have impairment of antioxidant defenses which are caused by a defect in activity of nuclear factor erythroid 2 like 2 (Nrf2), a prolific regulator of anti-oxidant enzymes, glutathione homeostasis, and cytoprotective proteins. Activation of Nrf2 protects mice with chronic smoke exposure from developing emphysema, decreases oxidative stress, increases proteasomal anti-apoptotic cytoprotective responses, improves bacterial phagocytosis and killing, and reverses tobacco-smoke induced corticosteroid resistance. Similarly, in vitro Nrf2 activation in human COPD lung cells has shown improved cytoprotection, improved bacterial clearance, and restoration of steroid sensitivity. This trial focuses on sulforaphane, a derivative of cruciferous vegetables, which is a potent in vitro and in vivo stimulator of Nrf2 activity. The investigators want to investigate whether ingestion of sulforaphane by chronic obstructive pulmonary disease (COPD) patients will increase Nrf2 activity and expression of downstream antioxidants in alveolar macrophages and bronchial epithelial cells. Accordingly, the investigators are conducting a placebo-controlled randomized proof of principle trial of two oral doses of sulforaphane, 25 and 150 micromoles, for 4 weeks in 90 COPD patients. Collections of alveolar macrophages by Bronchoalveolar lavage (BAL), bronchial epithelial cells by endobronchial brushings will be performed at baseline and 4 weeks. Other bio-specimens will include nasal epithelial cells, Peripheral Blood Monocyte Collection (PBMCs), and expired breath condensate (EBC). The investigators' goal is to establish a safe and tolerable dose of sulforaphane that effects in vivo antioxidants via Nrf2, then the investigators will have a novel candidate treatment for longer-term efficacy trials. Ancillary studies are proposed to explore the efficacy and mechanisms of sulforaphane to increase bacterial clearance and to restore steroid sensitivity in COPD lung cells.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or greater, either sex
* 10 or more pack-years smoking history
* Physician diagnosed COPD
* Post bronchodilator Forced expiratory volume in 1 second (FEV1)/ forced expiratory vital capacity (FVC) ratio < 0.70
* FEV1 40-80 % predicted
* Willingness to ingest no more than 1 serving of cruciferous vegetables per week during run-in and treatment periods
* Ability and willingness to provide informed consent

Exclusion Criteria:

* COPD exacerbation within preceding 6 weeks requiring treatment
* Significant respiratory (other than COPD), cardiovascular, neuropsychiatric, renal, gastrointestinal, or genitourinary disease that would interfere with participation in the study or interpretation of the results.
* Acute Myocardial infarction (MI) or Acute Coronary syndrome within 6 prior months
* Cancer (other than skin or localized prostate) within preceding 5 years
* Child-bearing potential with lack of adequate contraception, Pregnancy or lactation. Acceptable forms of birth control include abstinence, hysterectomy, tubal ligation, two of the following: vasectomy, condom, diaphragm, intrauterine device, oral or implanted contraceptives, or spermicide.
* Allergy to local anesthesia
* Resting hypoxemia (O2 saturation < 90%)
* Glomerular Filtration Rate (GFR) < 30
* Liver enzymes four times upper normal
* Current use of warfarin for any indication

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet T Holbrook, PhD, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (3):
- United States (3):
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - University at Baffalo, The State University of New York, Buffalo, New York
  - Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The primary method of data-sharing will be through the traditional mechanism of publication of results in the peer-reviewed medical literature. Following publication of the main results, in accordance with NIH policy, a de-identified, HIPAA-compliant limited use dataset will be made available to qualified investigators who have Institutional Review Board approval and sign a data-use agreement. De-identified specimens collected in the study that are not analyzed for the main study will be made available to qualified investigators along with a limited use dataset in line with University and Office of Human Research Protections guidelines with a materials transfer agreement and/or data-use agreement as applicable. The Center for Clinical Trials has extensive experience in preparation of limited use datasets, and maintains policies and model agreements for data-use agreements and materials-transfer agreements.

REFERENCES:
- [Derived] Sidhaye VK, Holbrook JT, Burke A, Sudini KR, Sethi S, Criner GJ, Fahey JW, Berenson CS, Jacobs MR, Thimmulappa R, Wise RA, Biswal S. Compartmentalization of anti-oxidant and anti-inflammatory gene expression in current and former smokers with COPD. Respir Res. 2019 Aug 20;20(1):190. doi: 10.1186/s12931-019-1164-1. PMID 31429757
- [Derived] Wise RA, Holbrook JT, Criner G, Sethi S, Rayapudi S, Sudini KR, Sugar EA, Burke A, Thimmulappa R, Singh A, Talalay P, Fahey JW, Berenson CS, Jacobs MR, Biswal S; Broccoli Sprout Extract Trial Research Group. Lack of Effect of Oral Sulforaphane Administration on Nrf2 Expression in COPD: A Randomized, Double-Blind, Placebo Controlled Trial. PLoS One. 2016 Nov 10;11(11):e0163716. doi: 10.1371/journal.pone.0163716. eCollection 2016. PMID 27832073

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Sulforaphane 25 | Sulforaphane 150
Started | 31 | 29 | 29
Completed | 29 | 28 | 28
Not Completed | 2 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Did not complete bronchoscopy | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sulforaphane 25 | Sulforaphane 150 | Total
Number analyzed (Participants) | 31 | 29 | 29 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 24 | 19 | 65
  >=65 years | 9 | 5 | 10 | 24
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [52 to 67] | 59 [54 to 65] | 56 [52 to 62] | 58 [54 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 8 | 35
  Male | 16 | 17 | 21 | 54
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 29 | 89
Chronic obstructive pulmonary disease (COPD) characteristics [Number; unit: participants]
  10 or more pack years of smoking history | 30 | 29 | 29 | 88
  Smoke cigarettes now | 20 | 16 | 18 | 54
  Smoke 10 or more cigarettes a day now | 10 | 9 | 10 | 29
  COPD exacerbation in last 12 months | 5 | 7 | 7 | 19
Post bronchodilator FEV1 [Median (Inter-Quartile Range); unit: percent predicted] — Forced expiratory volume in 1 second (FEV1) after administration of bronchodilator
  percent predicted | 61 [54 to 70] | 54 [50 to 65] | 65 [55 to 72] | 61 [53 to 70]
Post bronchodilator FEV1/FVC ratio [Median (Inter-Quartile Range); unit: ratio] — Ratio of forced expiratory volume in 1 second (FEV1) to forced vital capacity (FVC) after bronchodilation
  ratio | 0.56 [0.51 to 0.63] | 0.52 [0.47 to 0.59] | 0.57 [0.50 to 0.63] | 0.56 [0.48 to 0.62]
Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO) [Median (Inter-Quartile Range); unit: mL/mmHg/min] — DLCO: Diffusing capacity of the lungs for carbon monoxide measured by the single breath technique in accordance with American Thoracic Society standards
  mL/mmHg/min | 14.8 [11.8 to 19.5] | 15.7 [12.1 to 19.3] | 16.3 [12.3 to 21.4] | 15.7 [12.1 to 20.9]
Pulse oximetry (SpO2) [Median (Inter-Quartile Range); unit: Percentage of oxyhemoglobin] | 95 [94 to 97] | 96 [95 to 97] | 96 [94 to 97] | 96 [94 to 97]
Pulmonary function measures [Median (Inter-Quartile Range); unit: Liters] — Values were determined using either helium dilution or plethysmography methods, depending on equipment available at study sites. Lung volumes were measured in accordance with local hospital procedures.
  Liters
    Total lung capacity | 6.0 [4.7 to 7.3] | 5.5 [4.9 to 6.8] | 6.3 [5.7 to 7.0] | 6.0 [5.0 to 7.2]
    Slow vital capacity | 3.1 [2.4 to 4.1] | 3.0 [2.8 to 3.7] | 3.7 [3.1 to 4.4] | 3.3 [2.7 to 4.1]
    Forced residual capacity | 3.6 [3.1 to 4.5] | 3.6 [3.0 to 4.1] | 3.4 [3.0 to 3.9] | 3.5 [3.0 to 4.2]
    Residual volume | 2.6 [2.5 to 3.4] | 2.6 [2.2 to 3.5] | 2.7 [2.3 to 2.9] | 2.6 [2.2 to 3.2]
Use of respiratory medications in prior 2 weeks [Number; unit: participants]
  Short-acting beta-agonist | 22 | 21 | 18 | 61
  Long-acting beta-agonist | 2 | 1 | 2 | 5
  Long-acting beta-agonist & inhaled corticosteroid | 14 | 13 | 13 | 40
  Long-acting anticholinergic bronchodilator | 7 | 9 | 10 | 26
Medical Research Council Dyspnea Score [Median (Inter-Quartile Range); unit: units on a scale] — Minimum score 1, maximum score 5. Higher values represent a worse outcome.
  units on a scale | 2 [1 to 3] | 2 [2 to 3] | 2 [1 to 3] | 2 [1 to 3]
St Georges Respiratory Questionnaire [Median (Inter-Quartile Range); unit: units on a scale] — Scales, ranges, and descriptors:
  All scores are expressed as a percentage of overall impairment where 100 is the worst possible health status and 0 is the best possible health status.
  Total score (all items) summarizes the impact of the disease on overall health status Symptoms score (Q1-8) looks at the effect of respiratory symptoms, their frequency and severity.
  Activity score (Q11-17, 37-45) measures activities causing or limited by breathlessness Impacts score (Q18-36, 46-52) covers a range of aspects re: social functioning and psychological disturbances resulting from airways disease
  units on a scale
    Total score | 43 [24 to 58] | 47 [27 to 56] | 39 [24 to 54] | 40 [26 to 56]
    Symptoms score | 58 [32 to 70] | 55 [43 to 68] | 50 [31 to 57] | 52 [36 to 68]
    Activity score | 54 [30 to 74] | 60 [47 to 74] | 50 [41 to 73] | 55 [36 to 74]
    Impacts score | 27 [17 to 44] | 34 [15 to 46] | 26 [13 to 42] | 28 [15 to 44]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alveolar Macrophage Expression of Nrf2 and Associated Genes at 4 Weeks
Description: The first primary design variable is the change from baseline in nuclear factor erythroid 2 like 2 (Nrf2) expression in alveolar macrophages (AM) at 4 weeks by analysing Nrf2 protein and expression of a panel of Nrf2 regulated genes.Three participants - one from each treatment group - were unable to complete follow-up bronchoalveolar lavage for primary outcome data.
Time Frame: Baseline and 4 weeks
Population: Number of participants analyzed based on number of individuals with alveolar macrophage samples in which assays could be successfully performed. Assays failed for two participants in the placebo group, one in the 25 micromole group, and one in the 150 micromole group.
Measure: Median (Inter-Quartile Range); unit: fold change
Arm/Group | Placebo | Sulforaphane 25 | Sulforaphane 150
Number analyzed (Participants) | 27 | 27 | 27
fold change
  NQ01 | 0.80 [0.53 to 1.09] | 1.03 [0.56 to 1.60] | 0.94 [0.59 to 1.72]
  HO1 | 0.90 [0.69 to 1.34] | 0.98 [0.83 to 1.31] | 1.06 [0.68 to 1.74]
  AKR1C1 | 0.81 [0.46 to 1.27] | 1.13 [0.38 to 1.99] | 0.71 [0.56 to 1.57]
  AKR1C3 | 1.03 [0.76 to 1.37] | 1.02 [0.67 to 1.31] | 0.87 [0.40 to 1.32]
  Nrf2 | 1.14 [0.79 to 1.52] | 1.05 [0.87 to 1.47] | 1.13 [0.74 to 1.28]
  Keap1 | 0.94 [0.66 to 1.17] | 0.99 [0.82 to 1.11] | 1.06 [0.59 to 1.32]
Statistical Analysis 1: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Applies to gene expression of NAD(P)H Quinone Dehydrogenase 1 (NQ01) in alveolar macrophages; Test type: Superiority or Other; p = 0.45, Kruskal-Wallis
Statistical Analysis 2: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Applies to gene expression of Heme Oxygenase 1 (HO1) in alveolar macrophages; Test type: Superiority or Other; p = 0.40, Kruskal-Wallis
Statistical Analysis 3: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Applies to gene expression of Aldo-Keto Reductase Family 1 Member C1 (AKR1C1) in alveolar macrophages; Test type: Superiority or Other; p = 0.75, Kruskal-Wallis
Statistical Analysis 4: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Applies to gene expression of Aldo-Keto Reductase Family 1 Member C3 (AKR1C3) in alveolar macrophages; Test type: Superiority or Other; p = 0.49, Kruskal-Wallis
Statistical Analysis 5: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Applies to gene expression of nuclear factor erythroid 2 like 2 (Nrf2) in alveolar macrophages; Test type: Superiority or Other; p = 0.88, Kruskal-Wallis
Statistical Analysis 6: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Applies to gene expression of Kelch Like ECH Associated Protein 1 (Keap1) in alveolar macrophages; Test type: Superiority or Other; p = 0.71, Kruskal-Wallis

2. Primary Outcome: Change From Baseline in Bronchial Epithelial Cell Expression of Nrf2 at 4 Weeks
Description: The second primary design variable is the change from baseline in nuclear factor erythroid 2 like 2 (Nrf2) expression in bronchial epithelial cells (BEC) at 4 weeks by analysing Nrf2 protein. Three participants - one from each treatment group - were unable to complete follow-up bronchoalveolar lavage for primary outcome data.
Time Frame: Baseline and 4 weeks
Population: Number of participants analyzed based on number of individuals with bronchial epithelial samples in which assays could be successfully performed. Assays failed for one participant in the placebo group and one in the 25 micromole group..
Measure: Median (Inter-Quartile Range); unit: fold change
Arm/Group | Placebo | Sulforaphane 25 | Sulforaphane 150
Number analyzed (Participants) | 28 | 27 | 28
fold change | 1.09 [0.88 to 1.30] | 1.06 [0.92 to 1.28] | 1.06 [0.76 to 1.31]
Statistical Analysis 1: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Applies to gene expression of Nrf2 in bronchial epithelial cells; Test type: Superiority or Other; p = 0.68, Kruskal-Wallis

3. Primary Outcome: Change From Baseline in Bronchial Epithelial Cell Expression of NQ01 and Keap1 at 4 Weeks
Description: The third primary design variable is the change from baseline in NAD(P)H Quinone Dehydrogenase 1 (NQ01) and Kelch Like ECH Associated Protein 1 (Keap1) expression in bronchial epithelial cells (BEC) at 4 weeks. Three participants - one from each treatment group - were unable to complete follow-up bronchoalveolar lavage for primary outcome data.
Time Frame: Baseline and 4 weeks
Population: Number of participants analyzed based on number of individuals with bronchial epithelial samples in which assays could be successfully performed. Assays failed for two participants in the placebo group and one in the 150 micromole group.
Measure: Median (Inter-Quartile Range); unit: fold change
Arm/Group | Placebo | Sulforaphane 25 | Sulforaphane 150
Number analyzed (Participants) | 27 | 28 | 27
fold change
  NQ01 | 1.09 [0.83 to 1.50] | 1.12 [0.89 to 1.53] | 0.96 [0.65 to 1.41]
  KEAP1 | 1.12 [0.71 to 1.54] | 1.39 [0.99 to 2.24] | 0.87 [0.58 to 1.10]
Statistical Analysis 1: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Applies to gene expression of NAD(P)H Quinone Dehydrogenase 1 (NQ01) in bronchial epithelial cells; Test type: Superiority or Other; p = 0.69, Kruskal-Wallis
Statistical Analysis 2: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Applies to gene expression of Kelch Like ECH Associated Protein 1 (Keap1) in bronchial epithelial cells; Test type: Superiority or Other; p < 0.01, Kruskal-Wallis

4. Primary Outcome: Change From Baseline in Bronchial Epithelial Cell Expression of HO1 at 4 Weeks
Description: The fourth primary design variable is the change from baseline in expression of Heme Oxygenase 1 (HO1) in bronchial epithelial cells (BEC) at 4 weeks. Three participants - one from each treatment group - were unable to complete follow-up bronchoalveolar lavage for primary outcome data.
Time Frame: Baseline and 4 weeks
Population: Number of participants analyzed based on number of individuals with bronchial epithelial samples in which assays could be successfully performed. Assays failed for one participant in the placebo group.
Measure: Median (Inter-Quartile Range); unit: fold change
Arm/Group | Placebo | Sulforaphane 25 | Sulforaphane 150
Number analyzed (Participants) | 28 | 28 | 28
fold change | 1.05 [0.60 to 1.23] | 1.12 [0.82 to 1.67] | 0.93 [0.62 to 1.45]
Statistical Analysis 1: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Applies to gene expression of Heme Oxygenase 1 (HO1) in bronchial epithelial cells; Test type: Superiority or Other; p = 0.53, Kruskal-Wallis

5. Primary Outcome: Change From Baseline in Bronchial Epithelial Cell Expression of AKR1C1 at 4 Weeks
Description: The fifth primary design variable is the change from baseline in expression of Aldo-Keto Reductase Family 1 Member C1 (AKR1C1) in bronchial epithelial cells (BEC) at 4 weeks. Three participants - one from each treatment group - were unable to complete follow-up bronchoalveolar lavage for primary outcome data.
Time Frame: Baseline and 4 weeks
Population: Number of participants analyzed based on number of individuals with alveolar macrophage samples in which assays could be successfully performed. Assays failed for two participants in the placebo group and two in the 150 micromole group.
Measure: Median (Inter-Quartile Range); unit: fold change
Arm/Group | Placebo | Sulforaphane 25 | Sulforaphane 150
Number analyzed (Participants) | 27 | 28 | 27
fold change | 1.45 [0.84 to 1.98] | 1.08 [0.85 to 2.14] | 0.79 [0.53 to 1.08]
Statistical Analysis 1: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Applies to gene expression of Aldo-Keto Reductase Family 1 Member C1 (AKR1C1) in bronchial epithelial cells; Test type: Superiority or Other; p < 0.01, Kruskal-Wallis

6. Primary Outcome: Change From Baseline in Bronchial Epithelial Cell Expression of AKR1C3 at 4 Weeks
Description: The sixth primary design variable is the change from baseline in expression of Aldo-Keto Reductase Family 1 Member C3 (AKR1C3) in bronchial epithelial cells (BEC) at 4 weeks. Three participants - one from each treatment group - were unable to complete follow-up bronchoalveolar lavage for primary outcome data.
Time Frame: Baseline and 4 weeks
Population: Number of participants analyzed based on number of individuals with bronchial epithelial samples in which assays could be successfully performed. Assays failed for two participants in the placebo group, one participant in the 25 micromole group, and one participant in the 150 micromole group.
Measure: Median (Inter-Quartile Range); unit: fold change
Arm/Group | Placebo | Sulforaphane 25 | Sulforaphane 150
Number analyzed (Participants) | 27 | 27 | 27
fold change | 1.10 [0.74 to 1.62] | 1.38 [0.91 to 2.64] | 0.87 [0.50 to 1.68]
Statistical Analysis 1: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Applies to gene expression of Aldo-Keto Reductase Family 1 Member C3 (AKR1C3) in bronchial epithelial cells; Test type: Superiority or Other; p = 0.06, Kruskal-Wallis

7. Secondary Outcome: Fold-change in Isoprostane Concentrations (Follow-up to Baseline)
Description: Isoprostane, an oxidant stress indicator, was measured in expired breath condensate at baseline and 4 weeks.
Time Frame: Baseline and 4 weeks
Population: Number of participants analyzed based on number of individuals with expired breath condensate samples in which testing could be successfully performed. Samples were missing for two participants in the 25 micromole group and one participant in the 150 micromole group.
Measure: Median (Inter-Quartile Range); unit: fold change
Arm/Group | Placebo | Sulforaphane 25 | Sulforaphane 150
Number analyzed (Participants) | 30 | 27 | 28
fold change | 1.18 [0.42 to 1.79] | 0.83 [0.24 to 1.41] | 0.64 [0.29 to 1.33]
Statistical Analysis 1: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Test type: Superiority or Other; p = 0.20, Kruskal-Wallis

8. Secondary Outcome: Fold-change in Serum Inflammatory Marker Concentrations (Follow-up to Baseline)
Description: Inflammatory markers were measured in serum samples derived from venipuncture at baseline and 4 weeks in the serum of the participants of the trial.
Time Frame: Baseline and 4 weeks
Population: Number of participants analyzed is based on number of participants that had plasma samples available. Samples were missing for one participant in the 25 micromole group.
Measure: Median (Inter-Quartile Range); unit: fold change
Arm/Group | Placebo | Sulforaphane 25 | Sulforaphane 150
Number analyzed (Participants) | 30 | 28 | 29
fold change
  C-reactive protein (mg/L) | 0.99 [0.86 to 1.22] | 0.90 [0.69 to 1.06] | 1.01 [0.72 to 1.22]
  Interleukin-6 (pg/mL) | 0.75 [0.65 to 1.19] | 0.90 [0.76 to 1.08] | 1.12 [0.88 to 1.37]
  Interleukin-8 (pg/mL) | 1.06 [0.86 to 1.32] | 1.04 [0.87 to 1.17] | 1.03 [0.83 to 1.21]
Statistical Analysis 1: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Applies to C-reactive protein concentration; Test type: Superiority or Other; p = 0.41, Kruskal-Wallis
Statistical Analysis 2: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Applies to Interleukin-6 concentration; Test type: Superiority or Other; p = 0.07, Kruskal-Wallis
Statistical Analysis 3: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Applies to Interleukin-8 concentration; Test type: Superiority or Other; p = 0.65, Kruskal-Wallis

9. Secondary Outcome: Fold-change in Inflammatory Marker Concentrations in Bronchial Alveolar Lavage (Follow-up to Baseline) by Treatment Group
Description: Inflammatory markers were measured in bronchial alveolar lavage samples at baseline and 4 weeks in the participants of this trial who had bronchoalveolar lavage samples obtained.Three participants - one from each treatment group - were unable to complete follow-up bronchoalveolar lavage.
Time Frame: Baseline and 4 weeks
Population: Number of participants analyzed is based on number of participants that had bronchial alveolar lavage samples available. Samples were missing for two participants in the placebo group.
Measure: Median (Inter-Quartile Range); unit: fold change
Arm/Group | Placebo | Sulforaphane 25 | Sulforaphane 150
Number analyzed (Participants) | 27 | 28 | 28
fold change
  Interleukin-8 (pg/mg) | 1.22 [0.68 to 2.75] | 0.94 [0.52 to 2.22] | 1.11 [0.42 to 2.54]
  Secretory leukoprotease inhibitor (pg/mg) | 1.51 [0.83 to 1.90] | 1.09 [0.85 to 1.49] | 1.12 [0.65 to 1.51]
Statistical Analysis 1: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Applies to interleukin-8 results; Test type: Superiority or Other; p = 0.71, Kruskal-Wallis
Statistical Analysis 2: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Applies to secretory leukoprotease inhibitor results; Test type: Superiority or Other; p = 0.33, Kruskal-Wallis

10. Secondary Outcome: Fold-change in Plasma Inflammatory Marker Concentrations (Follow-up to Baseline)
Description: Inflammatory markers were measured in plasma at baseline and 4 weeks. Thiobarbituric acid reactive substances were measured in nmol malondialdehyde (MDA)/mL.
Time Frame: Baseline and 4 weeks
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: fold change
Arm/Group | Placebo | Sulforaphane 25 | Sulforaphane 150
Number analyzed (Participants) | 30 | 28 | 29
fold change
  Isoprostane (ng/mg) | 0.89 [0.55 to 1.22] | 0.90 [0.63 to 1.74] | 0.88 [0.55 to 1.37]
  Thiobarbituric acid reactive substances | 0.96 [0.77 to 1.19] | 1.05 [0.88 to 1.17] | 1.06 [0.84 to 1.27]
  Total antioxidants (mM Trolox equivalents/L) | 0.97 [0.92 to 1.03] | 0.92 [0.85 to 1.03] | 0.97 [0.90 to 1.04]
Statistical Analysis 1: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Applies to isoprostane results; Test type: Superiority or Other; p = 0.80, Kruskal-Wallis
Statistical Analysis 2: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Applies to thiobarbituric acid reactive substances results; Test type: Superiority or Other; p = 0.35, Kruskal-Wallis
Statistical Analysis 3: Comparison: Placebo vs Sulforaphane 25 vs Sulforaphane 150; Applies to total antioxidants results; Test type: Superiority or Other; p = 0.53, Kruskal-Wallis

ADVERSE EVENTS:
Description: Assessed via study questionnaires.
Arm/Group | Placebo | Sulforaphane 25 | Sulforaphane 150
Serious Adverse Events (participants affected / at risk) | 0/31 | 2/29 | 1/29
Other Adverse Events (participants affected / at risk) | 15/31 | 21/29 | 18/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=31) | Sulforaphane 25 (N=29) | Sulforaphane 150 (N=29)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=31) | Sulforaphane 25 (N=29) | Sulforaphane 150 (N=29)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 6 (6)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Poor appetite (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Bad taste in mouth (Gastrointestinal disorders) | 2 (2) | 7 (7) | 9 (9)
Heartburn (Gastrointestinal disorders) | 1 (1) | 6 (6) | 7 (7)
Headache (General disorders) | 2 (2) | 2 (2) | 1 (1)
Fatigue (General disorders) | 3 (3) | 5 (5) | 2 (2)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Bloating/gas (Gastrointestinal disorders) | 5 (5) | 7 (7) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 3 (3) | 6 (6)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Increased phlegm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No